CLINICAL TRIAL: NCT04950842
Title: Phase I/II Study to Evaluate the Safety and Efficacy of JB-101(Induced T Cell With Suppressing Functions), to Induce Operational Tolerance in Living Donor Liver Transplantation.
Brief Title: Induction of Transplant Tolerance in LDLT Via iTS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Juntendo University (Other)
Collaborators: Junten Bio Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Koichiro Uchida, Associate Professpr, Juntendo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jRCT2073200067
Record Dates: First submitted 2021-04-09; First posted 2021-07-06 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Living-donor Liver Transplantation
Keywords: living-donor liver transplantation; immunotolerance; operational tolerance; cell therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JB-101 (Experimental): induced T cell with suppressive function
  Interventions: Biological: JB-101

INTERVENTIONS:
Biological: JB-101 — induced T cell with suppressive function

SUMMARY:
The purpose of this clinical trial is to examine the immunotolerance-inducing ability (effectiveness) of induced inhibitory T cells JB-101 in patients with living-donor liver transplantation using "whether or not operational tolerance is achieved" as an index.

And the safety of JB-101 will be evaluated.

DETAILED DESCRIPTION:
This trial is a phase I / II, open-label, single-arm, multicenter clinical trial of JB-101, an inducible inhibitory T cell, in patients with end-stage liver failure who undergo living-donor liver transplantation.

The primary endpoint of efficacy is withdrawal from immunosuppressant by 78 weeks (up to 91 weeks) after liver transplantation, and then "whether or not operational tolerance is achieved".

ELIGIBILITY:
Inclusion Criteria：

Patients with end-stage liver failure undergoing living-donor liver transplantation.

Subjects who are healthy physically and psychologically and willing to donate organs voluntarily.

Relative within the second degree of relationship or partner. (Acceptable degree conforms eligibility criteria of the institution.)

Exclusion Criteria：

Patients who have clinical findings of active infection.

Patients with advanced heart disease, fulminant hepatitis in liver failure, renal disease, malignant tumors and complications of immunodeficiency.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Achievement of operational tolerance | immunosuppressive drug cessation was maintained for at least 12 months
  Achievement of "Operational Tolerance" defined as no biopsy proven rejection diagnosed by Banff criteria for more than 52 weeks after withdrawal of immunosuppressive drugs post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Koichiro Uchida, M.D.,Ph.D., Study Chair — Juntendo University Advanced Research Institute for Health Science
Locations (5):
- Japan (5):
  - Juntendo University Hospital, Bunkyoku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Kyoto University Hospital, Kyoto
  - Nagasaki University Hospital, Nagasaki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Todo S, Yamashita K, Goto R, Zaitsu M, Nagatsu A, Oura T, Watanabe M, Aoyagi T, Suzuki T, Shimamura T, Kamiyama T, Sato N, Sugita J, Hatanaka K, Bashuda H, Habu S, Demetris AJ, Okumura K. A pilot study of operational tolerance with a regulatory T-cell-based cell therapy in living donor liver transplantation. Hepatology. 2016 Aug;64(2):632-43. doi: 10.1002/hep.28459. Epub 2016 Mar 10. PMID 26773713